CLINICAL TRIAL: NCT05864261
Title: A Randomized, Blinding, Single-dose, Positive-drug Parallel Control Study to Compare the Pharmacokinetics Following Administration of JT1801 and Darbepoetin Alfa Injection (NESP®) in Chinese Healthy Adult Volunteers
Brief Title: Pharmacokinetics Comparison Study of JT1801 and NESP® After Single Dose Administration in Chinese Health Male Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yi Fang (Other)
Responsible Party: Sponsor-Investigator, Yi Fang, Professor of Pharmacy, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-I-JT1801-01
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Renal Anemia
MeSH Terms: interventions — Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JT1801 (Experimental)
  Interventions: Drug: JT1801 60ug
- NESP (Active Comparator)
  Interventions: Drug: NESP 60ug

INTERVENTIONS:
Drug: JT1801 60ug — JT1801, 60ug, IV injection
  Arms: JT1801
Drug: NESP 60ug — NESP, 60ug, IV injection
  Arms: NESP

SUMMARY:
The purpose of this study is to compare the similarity of major pharmacokinetic parameters after a single intravenous administration of JT1801 and NESP® in chinese healthy male volunteers. And to evaluate the safety, immunogenicity and pharmacodynamic characteristics of JT1801 and NESP® in chinese healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Chinese healthy adult male subjects.
2. Age of 18 to 55 years, inclusive.
3. Subject with BMI between 19 kg/m2 and 26 kg/m2 (inclusive); and a total body weight ≥50 kg.
4. Subject who agree to practive effective barrier contraception and avoid sperm donation during the entire study period and through at least 3 months after the last dose of study drug.
5. Subject who provided written informed consent voluntarily after being fully informed of the study.
6. Subject who is able to communicate well with the investigator and participate in the whole study process according to protocol.

Exclusion Criteria:

1. During the screening period, vital signs measurement, physical examination, laboratory examination (blood routine, reticulocyte, urine routine, blood biochemistry, coagulation function, anemia, transferrin saturation, IgE detection), B-ultrasound examination, chest X-ray and 12-lead electrocardiogram examination showed abnormal results and were judged by the investigator to be clinically significant.
2. History of chronic disease or serious disease in cardiovascular, liver, kidney, biliary tract, respiratory, blood, lymphatic, endocrinological, immunologic, psychiatric, neuromuscular, gastrointestinal system within three years.
3. Have a history of specific allergies (e.g. hives) or are allergic (e.g. are known to be allergic to two or more drugs), or have a history of allergy to this ingredient or to EPO drugs.
4. Subjects with past or present history of hypertension, stroke, thromboembolism, convulsion, epilepsy or pure red cell aplasia.
5. Subject with severe psychological or mental illness.
6. Subject with a previous history of tumors.
7. The investigator considers that there are other medical conditions that may affect the study results and the safety of the subjects.
8. Subject who had surgery within 6 months prior to screening period that the investigators determined would affect drug absorption, distribution, metabolism, or excretion, or who planned to have surgery during the study period.
9. Subject who have received other biologics within 6 months.
10. Those with a history of drug abuse (including the use of various narcotic drugs and psychotropic substances for non-medical destinations) or positive drug abuse screening (including morphine, methamphetamine, ketamine, dimethylenedioxyamphetamine, tetrahydrocannabinolic acid, etc.) before the test.
11. Positive for any of the virological tests, including human immunodeficiency virus, hepatitis C antibody, hepatitis B surface antigen, and treponema pallidum antibody.
12. Subjects who have donated blood or lost blood from other reasons within 6 months prior to screening with a total of 400mL or received blood transfusions or used blood products.
13. Has a history of alcohol abuse within 1 year prior to screening, whereby drink more than 2 units of alcohol per week on average (1 unit =360 mL beer or 45 mL liquor with 40% alcohol or 150 mL wine), or alcohol breath test results greater than 0.0mg/100 ml.
14. In the past year, the average daily consumption of excessive tea, coffee and/or caffeinated beverages (more than 8 cups, 1 cup ≈250mL).
15. Those who smoked > 5 cigarettes per day within 3 months before screening or could not refrain from smoking during the test.
16. Those who have used any drugs (prescription drugs, over-the-counter drugs, vitamins, Chinese herbal medicines, health supplements) within 30 days before enrollment.
17. Those who have used systemic glucocorticoids within 3 months before enrollment.
18. Those who have participated in other clinical trials within 3 months before enrollment.
19. Those who cannot tolerate venipuncture or have a history of needle sickness and blood sickness.
20. Those who have special requirements for diet and cannot accept a unified diet.
21. Subjects who received the vaccine within 3 months prior to the first dosing, or plan to be vaccinated during the study or within 1 week after the last dosing.
22. Those with a low probability of enrollment or poor adherence (such as frailty, physical exhaustion, dehydration or malnutrition, etc.) according to the judgment of the investigator.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 74 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
AUC0-t | Pre-dose and after dose 20 days
  PK parameters comparison between JT1801 and darbepoetin alfa: AUC0-t
AUC0-∞ | Pre-dose and after dose 20 days
  PK parameters comparison between JT1801 and darbepoetin alfa: AUC0-∞

SECONDARY OUTCOMES:
TEmax | Pre-dose and after dose 15 days
  PD parameters comparison between JT1801 and darbepoetin alfa: TEmax of reticulocyte count, hematocrit, hemoglobin concentration, RBC
Emax | Pre-dose and after dose 15 days
  PD parameters comparison between JT1801 and darbepoetin alfa: Emax of reticulocyte count, hematocrit, hemoglobin concentration, RBC
AUEC0-t | Pre-dose and after dose 15 days
  PD parameters comparison between JT1801 and darbepoetin alfa: AUEC0-t of reticulocyte count, hematocrit, hemoglobin concentration, RBC
ΔAUEC0-t | Pre-dose and after dose 15 days
  PD parameters comparison between JT1801 and darbepoetin alfa: ΔAUEC0-t of reticulocyte count, hematocrit, hemoglobin concentration, RBC
ΔEmax | Pre-dose and after dose 15 days
  PD parameters comparison between JT1801 and darbepoetin alfa: ΔEmax of reticulocyte count, hematocrit, hemoglobin concentration, RBC

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No